CLINICAL TRIAL: NCT04663529
Title: Correlation Study of Corneal Nerve Changes and Dry Eye in Contact Lens Wearers
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CLADE
Record Dates: First submitted 2020-09-16; First posted 2020-12-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2020-09

CONDITIONS: Contact Lens Complication; Dry Eye
Keywords: contact lens; tear film; dry eye; corneal sub-basal nerve
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Contact Lenses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tear
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CLADE: contact lens wearers with DED
  Interventions: Other: contact lens
- non-CLADE: DED without contact lens wear
- NC: normal control

INTERVENTIONS:
Other: contact lens — daily disposable soft contact lens
  Groups: CLADE

SUMMARY:
This study aims to analyze the changes of corneal nerve morphology and function in contact lens-related dry eye(CLADE) patients and further discuss the role of corneal nerve in the genesis and development of CLADE.

DETAILED DESCRIPTION:
33 daily disposable soft contact lens wearers with dry eye disease(DED), 33 DED without contact lens wear and 33 normal control subjects will be involved in study. One experienced ophthalmologist will evaluate the DED symptoms and signs, which include ocular surface disease index(OSDI), tear film breakup time(TBUT), Schirmer Ⅰ test, corneal fluorescein staining, lissamine green staining and meibomian gland dropout rate. After evaluating, corneal sensitivity are measured using a Cochet-Bonnet aesthesiometer. Corneal nerve morphology will be assessed in the right eye using in vivo confocal microscopy(IVCM). Fifteen to twenty minutes after IVCM, 20μL of basal tears will be collected from the inferior meniscus of each participant to test tear neuropeptides. Then investigators analyse the correlation of corneal nerve changes and DED symptoms and signs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18years to 40 years；
* Male or female DED patients based on Chinese Dry Eye Diagnosis Standard (2020) with or without contact lens wear；
* Provision of written informed consent.

Exclusion Criteria:

* Presence of any of the following conditions: active ocular infection, ocular inflammation, active ocular allergy, ocular surgical history, laser treatment in the last 3 months, Meibomian function (MGD) over grade 2 (the grade is according to the report of the International Workshop on MGD in 2011), severe blepharitis or obvious inflammation of the eyelid margin, which in the judgment of the investigator may interfere with the interpretation of the study results
* Pregnant and lactating women, or those planning a pregnancy over the course of the study
* Uncontrolled systemic disease
* Suffer from diseases that may affect corneal nerves, such as keratoconus, trigeminal neuralgia, allergic conjunctivitis, etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: DED patients from Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
sub-basal corneal nerve density | baseline
  Sub-basal corneal nerve plexus image will be acquired using a laser scanning confocal microscope. Sub-basal nerve fiber density will be calculated from a manual trace of the length of all nerve fibers in each 1 mm2 image.
sub-basal corneal nerve tortuosity | baseline
  Sub-basal corneal nerve plexus image will be acquired using a laser scanning confocal microscope. Sub-basal nerve tortuosity will be assessed using a grading scale separately by two experienced ophthamologist.

SECONDARY OUTCOMES:
ocular surface disease index(OSDI) | baseline
  OSDI is one of the most frequently used questionnaires for evaluation of DED. This includes 12 questions which measure the frequency of symptoms over the recent week, and the scores range from 0 to 100.
Tear break-up time (TBUT) | baseline
  TBUT is the time from normal blinking to the first appearance of a break in the tear film.
Schirmer Ⅰ test (SⅠt) | baseline
  The Schirmer I test is performed using sterile strips without anesthesia. The strips are placed in the lateral part of the inferior fornix of the eye for 5min and the extent of tear flow down was measured in millimeters.
Corneal fluorescein staining | baseline
  The degree of fluorescein staining of the cornea was evaluated using the National Eye Institute (NEI) scale of five corneal regions (central, superior, temporal, nasal, and inferior).
Lissamine green staning | baseline
  To grade the temporal zone, the subject looks nasally; to grade the nasal zone the subject looks temporally. The upper and lower conjunctiva can also be graded.
meibomian gland droupout rate | baseline
  meibomian gland evaluation
corneal sensitivity | baseline
  Corneal sensitivity will be measured in the right eye only using the Cochet-Bonnet aesthesiometer and the ascending method of limits to determine the threshold of stimulus detection.
the concentration of substance P | baseline
  20μL of basal tears will be collected from the inferior meniscus of each subject to test substance P. Substance P levels will be quantified by competitive enzyme-linked immunosorbent assays.
the concentration of CGRP | baseline
  CGRP levels will be quantified by competitive enzyme-linked immunosorbent assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China